CLINICAL TRIAL: NCT02848885
Title: The Clinical and Functional Imaging Effects of Transcranial Direct Current Stimulation (tDCS) on Illness Awareness in Schizophrenia
Brief Title: The Effects of tDCS on Illness Awareness in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Philip Gerretsen, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 043-2016
Record Dates: First submitted 2016-07-15; First posted 2016-07-29 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Schizophrenia
Keywords: Magnetic resonance imaging; Anosognosia; Electrical stimulation of the brain
MeSH Terms: conditions — Schizophrenia; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active TDCS (Experimental): Participants who are randomly assigned to this arm will receive dual hemisphere parietal (P3 cathodal, P4 anodal) stimulation daily for 10 days. Each participant will have two MRI scans and their degree of illness awareness assessed at baseline and after 10 days of tDCS. Illness awareness will be assessed weekly thereafter for 4 weeks.
  Interventions: Other: Active TDCS
- Sham TDCS (Experimental): Participants who are randomly assigned to this arm will receive dual hemisphere sham stimulation with electrodes placed on the parietal lobes (P3 and P4) daily for 10 days. Each participant will have two MRI scans and their degree of illness awareness assessed at baseline and after 10 days of tDCS. Illness awareness will be assessed weekly thereafter for 4 weeks.
  Interventions: Other: Sham TDCS

INTERVENTIONS:
Other: Active TDCS — Participants will receive active tDCS stimulation.
  Arms: Active TDCS
Other: Sham TDCS — Participants will receive sham tDCS stimulation
  Arms: Sham TDCS

SUMMARY:
This is a novel study that seeks to explore the clinical and functional imaging effects of transcranial direct current stimulation (tDCS) on illness awareness or anosognosia in schizophrenia, arguably the most treatment-resistant manifestation of the disorder.

DETAILED DESCRIPTION:
Transcranial DCS is a novel, non-invasive and non-convulsive technique for altering brain function. To our knowledge, no research has investigated the functional and behavioural effects of tDCS on anosognosia in schizophrenia. As such, we aim to improve impaired illness awareness in schizophrenia with tDCS by inhibiting left hemisphere regions (i.e. temporoparietooccipital cortex) shown by our group to be activated during illness denial.

Positive results will demonstrate that impaired illness awareness in schizophrenia involves a similar brain network to impaired illness awareness in patients with brain lesions and can be similarly modulated with non-invasive techniques, such as tDCS. If proven effective, this easy to administer, safe, non-invasive intervention would have the potential to alter individuals' attitude towards their illness and medication, leading ultimately to an improvement in individuals' capacity for illness recognition and treatment engagement, which would undoubtedly have a significant impact on the management of this devastating mental disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female inpatients or outpatients ≥ 18 years of age
2. Having a DSM-IV diagnosis of schizophrenia or schizoaffective disorder
3. Voluntary and capable of consenting to participation in the research study
4. Fluent in English
5. Moderate-to-severe lack of illness awareness (≥3 on PANSS G12 Insight and Judgment item)
6. On a stable dose of antipsychotic and other concomitant medications, and unlikely to undergo changes in dose during the study

Exclusion Criteria:

1. Serious unstable medical illness or any concomitant major medical or neurological illness, including a history of seizures or a first degree relative with a history of a seizure disorder
2. Acute suicidal and/or homicidal ideation
3. Formal thought disorder rating of over 2 on the (Scale for Assessment of Positive Symptoms) SAPS.
4. DSM-IV substance dependence (except caffeine and nicotine) within one month prior to entering the study
5. Pregnant women
6. Mild lack of insight to good illness awareness (<3 on PANSS G12 Insight and Judgment item).
7. Positive urine drug screen for drugs of abuse
8. Currently taking antiepileptics
9. Any contraindications to MRI (eg., metal implants that would preclude an MRI, claustrophobia)
10. Score < 32 on the Wide Range Achievement Test-III (WRAT III)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Illness awareness | At baseline and weekly for 4 weeks after tDCS
  The primary aim of this study is to determine if dual hemisphere tDCS daily for 10 days will lead to an improvement in illness awareness versus a control condition (sham tDCS), as measured by changes in illness awareness scores post intervention (10 days post tDCS and weekly x 4 weeks post tDCS) in participants with schizophrenia.

SECONDARY OUTCOMES:
Neural activity | At baseline and post TDCS
  A secondary aim of this study is to assess changes in brain network activity (blood oxygen level dependent-BOLD) before and after tDCS while performing an illness awareness task during functional MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gerretsen, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.net/research